CLINICAL TRIAL: NCT05662371
Title: Influence of Nociception Level Monitor (NOL) Guided Analgesic Delivery on the Perioperative Course, Quality of Recovery and Hospital Stay in Robot-assisted Colorectal Surgery
Brief Title: Influence of Nociception Level Monitor (NOL) Guided Analgesic Delivery on Robot-assisted Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHS-An-3-2022
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use, Unspecified; Pain, Postoperative
Keywords: Nociception,; robotic surgery,; opioids,; postoperative recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Clinical Care Group (Placebo Comparator): Hemodynamic changes outside of the normal range i.e., hypertension (systolic blood pressure greater than 140 mm Hg), tachycardia (heart rate greater than 90 min-1) and hypotension (mean arterial pressure less than 60 mm Hg) will be first assessed using the guidance of Bispectral index and Train of four monitors. Sufentanil in doses of 2.5 to 5 mcg (maximum of 0.6-1.2 mic/kg for the entire surgery) is administered if the Bispectral index and Train of four monitor values are within normal range and if required vasopressor infusion is used. Vasoconstrictors may be given as a continuous infusion of norepinephrine, or bolus doses of ephedrine or phenylephrine. Only when blood pressure remains, low additional crystalloids will be given. Finally, in case of bradycardia (heart rate less than 30 min-1), atropine may be given
  Interventions: Device: Standard care
- Nociception Level-guided Analgesia Group (Experimental): In the nociception level-guided group, sufentanil will be administered to maintain a nociception level value between 10 and 25. In case the nociception level values rise greater than 25 for more than 60 s, additional 2.5 microgram sufentanil (if nociception level increase remained less than 45) or 5 micrograms (if nociception level increase greater than 45). Atropine will be administered when heart rate decreases less than 30 min-1. Because the nociception level may be sensitive to such medication, nociception level values will then not used for at least 5 min to guide analgesia, with the exception of norepinephrine as this drug will be given as continuous infusion
  Interventions: Device: Nociception Level monitor (NOL)

INTERVENTIONS:
Device: Nociception Level monitor (NOL) — NOL technology uses a multiparameter-based sensor platform, and advanced algorithm, to continuously monitor Autonomic Nervous System (ANS) functions. NOL reflects a patient's nociceptive state and analgesic effect, helping to optimize the administration of systemic and/or regional analgesics, and avoiding overdose or underuse of these drugs. The nociception level is a multiparameter monitor that combines information from the finger photoplethysmogram amplitude, skin conductance, skin conductance fluctuation, heart rate, heart rate variability, and their time derivatives into one index ranging from 0 (absence of noxious stimulation) to 100 (severe noxious stimulation).
  Arms: Nociception Level-guided Analgesia Group
Device: Standard care — Hemodynamic changes outside of the normal range i.e., hypertension (systolic blood pressure greater than 140 mm Hg), tachycardia (heart rate greater than 90 min-1) and hypotension (mean arterial pressure less than 60 mm Hg) will be first assessed using the guidance of Bispectral index and Train of four monitors. Sufentanil in doses of 2.5 to 5 mcg (maximum of 0.6-1.2 mic/kg for the entire surgery) is administered if the Bispectral index and Train of four monitor values are within normal range and if required vasopressor infusion is used. Vasoconstrictors may be given as a continuous infusion of norepinephrine, or bolus doses of ephedrine or phenylephrine. Only when blood pressure remains, low additional crystalloids will be given. Finally, in case of bradycardia (heart rate less than 30 min-1), atropine may be given
  Arms: Standard Clinical Care Group

SUMMARY:
Being relatively new, the NOL monitor may offer interesting observations in perioperative nociception levels and appropriate analgesic consumption in diverse surgeries, including robot-assisted surgery. These observations may supplement the current efforts towards further advantages in rapid restitution. Therefore, the investigators planned a trial where intra-operative analgesics were guided using an NOL monitor to study if intra-operative NOL guidance influences peri-operative analgesic consumption, postoperative length of stay and quality of recovery of patients subjected for robot-assisted surgery.

DETAILED DESCRIPTION:
During anesthesia for surgical procedures, anesthetic and muscle relaxant drugs can be meticulously administered using Bispectral Index (BIS) and neuromuscular monitors. However, analgesic drugs are still dispensed using poor surrogate parameters such as heart rate and blood pressure. This subjective dosing of analgesic drugs may invariably lead to inappropriate intra-operative consumption. This may result in tachycardia, hypertension, and postoperative pain due to e.g. insufficient analgesia, or hypotension, bradycardia, respiratory depression and Post-Operative Nausea and Vomiting (PONV) secondary to excessive analgesia. These effects may be detrimental to the patients especially those with multiple comorbidities with limited vital organ reserves such as patients classified to III or IV by the American Society of Anaesthesia classification (ASA) Similarly, immediate postoperative recovery may also get delayed due to pain, unstable hemodynamics, nausea and vomiting. In that context, there has long been search for a monitor which can guide meticulous administration of analgesics. Recently, a Nociception Level monitor (NOL) based on advanced software algorithms using multiple physiological parameters has been developed. It offers an objective score (NOL Index) which relates to the level of intra-operative pain. NOL technology has been validated and found superior to existing pain indicators in peer-reviewed publications. The NOL monitor may offer interesting observations in perioperative nociception levels and appropriate analgesic consumption in diverse surgeries, including robot-assisted surgery. These observations may supplement the current efforts towards further advantages in rapid restitution. Therefore, the investigators are planning a trial where intra-operative analgesics are guided using an NOL monitor.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists score III-IV
* Scheduled for elective major robot-assisted colorectal surgeries

Exclusion Criteria:

* Inability to give informed consent
* planned spinal or epidural anaesthesia
* all forms of regional anaesthesia, including wound infiltration
* nonelective procedures
* pregnancy or lactation
* atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total intraoperative consumption of sufentanil Total intraoperative consumption of sufentanil | From induction of anaesthesia up to transfer to recovery room, up to 6 hours
  Amount of sufentanil in micrograms administered during the entire operative period i.e. from induction of anaesthesia up to transfer to the recovery room

SECONDARY OUTCOMES:
Eligible time to discharge as per RR discharge score | From admission to recovery room until discharge, up to 24 hours
  The RR discharge score is a scoring system developed for general surgery by the Danish Society of Anesthesia and Intensive Care. The score consists of 5 semi-objective variables (sedation, respiration, nausea, pain, and motor function) and 5 objective variables (peripheral saturation, diuresis, arterial blood pressure, heart rate and temperature). The nurses score each variable from 0 to 3 points. Low scores( below 3 for 2 consecutive hours) indicate a stable condition, and patients are considered eligible for discharge. The score values at different time points represent the quality of recovery.
Postoperative Nausea and Vomiting | From admission to recovery room, up to 24 hours
  Complaint from patient about nausea on arrival in recovery room assessed as yes or no
Change in myocardial function | Before anaesthesia induction and 24 hours after completion of surgery
  Difference between preoperative and postoperative (24 hours after surgery) Serum Troponin T and brain natriuretic peptide (proPnP) levels

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Strøm, Study Director — Hospital of Southern Denmark - Aabenraa
Locations (1):
- Anaesthesiology and Intensive Care Research Unit, Aabenraa, Denmark